CLINICAL TRIAL: NCT01842815
Title: Evaluation of the 755nm Alexandrite for Unwanted Tattoos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PICO-SK
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Unwanted, Non Cosmetic, Tattoos
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 755nm Alexandrite Laser Single Pass (Right Side). (Experimental): 755nm Alexandrite Laser for Treatment of unwanted, non cosmetic tattoos. The right side will be treated once within the same visit.
  Interventions: Device: 755 nm alexandrite laser
- 755nm Alexandrite Laser Double Pass (Left Side) (Experimental): 755nm Alexandrite Laser for Treatment of unwanted, non cosmetic tattoos. The left side of the tattoo will be treated twice within the same visit 20 minutes apart.
  Interventions: Device: 755 nm alexandrite laser

INTERVENTIONS:
Device: 755 nm alexandrite laser — 755 nm alexandrite laser for the treatment of unwanted, non cosmetic, tattoos.

SUMMARY:
The purpose of this study is to collect further data on the safety and efficacy of removing unwanted non cosmetic tattoos (including recalcitrant) using a 755nm Alexandrite laser.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 85 years old.
2. Has unwanted non-cosmetic tattoo(s) and wishes to undergo laser treatments to remove them.
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria:

1. Is hypersensitive to light exposure.
2. Has active localized or systemic infection.
3. Is taking medication(s) for which sunlight is a contraindication.
4. Has a history of squamous cell carcinoma or melanoma.
5. Has a history of keloid scarring.
6. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment.
7. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
8. Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
9. Is allergic to lidocaine, tetracaine or Xylocaine with epinephrine.
10. Has any other reason determined by the physician to be ineligible to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Laser & Skin Surgery Center of Northern California, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects are enrolled in both study arms because all subjects will be receiving treatment on the left side of the tattoo and treatment on the right side of the tattoo in each visit.
Units Other Than Participants: treatment areas
Groups:
- 755nm Alexandrite Laser: 755nm Alexandrite Laser for Treatment of unwanted, non cosmetic tattoos
  755 nm alexandrite laser: 755 nm alexandrite laser for the treatment of unwanted, non cosmetic, tattoos.
Period: Overall Study
Arm/Group | 755nm Alexandrite Laser
Started | 20; 26 treatment areas
Completed | 16; 22 treatment areas
Not Completed | 4; 4 treatment areas

BASELINE CHARACTERISTICS:
Population: 1 subject withdrew, per sponsor request, due to multiple laser devices already used on treatment area. They withdrew before baseline information was taken of them.
Arm/Group | 755nm Alexandrite Laser
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 12
  Race/Ethnicity: Asian | 0
  Race/Ethnicity: African American | 1
  Race/Ethnicity: Hispanic | 4
  Race/Ethnicity: Native American | 1
  Race/Ethnicity: Other | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 1
    Fitzpatrick Skin Type II | 6
    Fitzpatrick Skin Type III | 7
    Fitzpatrick Skin Type IV | 4
    Fitzpatrick Skin Type V | 1
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Clearance
Description: Clearance will be measured using a clearance aesthetic improvement scale. This scale ranges from 0 to 10, where 0 is 0% tattoo cleared compared to the baseline tattoo, and 10 is 100% of tattoo cleared compared to the baseline tattoo.
Time Frame: Post Treatment 1 (6 Weeks Post Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: tattoos
Arm/Group | 755nm Alexandrite Laser Single Pass (Right Side). | 755nm Alexandrite Laser Double Pass (Left Side)
Number analyzed (Participants) | 19 | 19
Number analyzed (tattoos) | 24 | 24
score on a scale | 2.875 (2.112) | 4.25 (2.513)
Statistical Analysis 1: Comparison: 755nm Alexandrite Laser Single Pass (Right Side). vs 755nm Alexandrite Laser Double Pass (Left Side); This t-test is to test the statistical significance of the right side of the tattoo clearance vs. the left side of the tattoo clearance. It tests if there is a difference between the tattoo being treated twice per visit (right side) vs. being treated once per visit (left side); Test type: Superiority; p = .0077, t-test, 2 sided — The value looked at for statistical significance is if p<.05; t-tailed, paired t-test

2. Primary Outcome: Tattoo Clearance
Description: as for outcome 1
Time Frame: Post Treatment 2 (12 Weeks Post Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: tattoos
Arm/Group | 755nm Alexandrite Laser Single Pass (Right Side). | 755nm Alexandrite Laser Double Pass (Left Side)
Number analyzed (Participants) | 19 | 19
Number analyzed (tattoos) | 24 | 24
score on a scale | 3.75 (2.21) | 4.88 (2.58)
Statistical Analysis 1: Comparison: 755nm Alexandrite Laser Single Pass (Right Side). vs 755nm Alexandrite Laser Double Pass (Left Side); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .00012, t-test, 2 sided — The value looked at for statistical significance is if p<.05; t-tailed, paired t-test

3. Primary Outcome: Tattoo Clearance
Description: as for outcome 1
Time Frame: Post Treatment 3 (18 Weeks Post Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: tattoos
Arm/Group | 755nm Alexandrite Laser Single Pass (Right Side). | 755nm Alexandrite Laser Double Pass (Left Side)
Number analyzed (Participants) | 19 | 19
Number analyzed (tattoos) | 24 | 24
score on a scale | 4.5 (2.48) | 5.77 (2.83)
Statistical Analysis 1: Comparison: 755nm Alexandrite Laser Single Pass (Right Side). vs 755nm Alexandrite Laser Double Pass (Left Side); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .0034, t-test, 2 sided — The value looked at for statistical significance is if p<.05; t-tailed, paired t-test

ADVERSE EVENTS:
Time Frame: Adverse data were collected from the first treatment until 3 months post-treatment.
Description: The adverse events were reported in 1 group instead of 2 (right vs. left) because that distinction in adverse events collection was not examined or required for this study's aims.
Arm/Group | 755nm Alexandrite Laser
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 755nm Alexandrite Laser (N=20)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Blistering (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.